CLINICAL TRIAL: NCT01047202
Title: A Blinded, Randomized and Controlled Clinical Trial With Influenza A/H1N1 Split-virion Vaccine in 6 to 35 Months Infants
Brief Title: Sinovac, Pandemic Influenza A/H1N1 Vaccine in 6 to 35 Months Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-PanFlu-4003
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (3):
- Group 1: 7.5 μg pandemic influenza A/H1N1 vaccine (Experimental): 120 subjects to receive two doses of 7.5 μg pandemic influenza A/H1N1 vaccine 21 days apart
  Interventions: Biological: Pandemic influenza A/H1N1 vaccine
- Group 2 : 15 μg pandemic influenza A/H1N1 vaccine (Experimental): 120 subjects to receive two doses of 15 μg pandemic influenza A/H1N1 vaccine 21 days apart
  Interventions: Biological: Pandemic influenza A/H1N1 vaccine
- Group 3 : 7.5 μg seasonal trivalent vaccine (Sham Comparator): 60 subjects to receive two doses of 7.5 μg seasonal trivalent vaccine 21 days apart
  Interventions: Biological: Seasonal trivalent vaccine

INTERVENTIONS:
Biological: Pandemic influenza A/H1N1 vaccine — Pandemic influenza A/H1N1 vaccine (PANFLU.1), 15 micrograms per dose per 0.5 millilitre. Vaccines will be administered as a single 0.25 mL intramuscular injection in the deltoid muscle of the arm (randomized in one arm) at the first dose and the other arm for the second dose
  Arms: Group 1: 7.5 μg pandemic influenza A/H1N1 vaccine
Biological: Pandemic influenza A/H1N1 vaccine — Pandemic influenza A/H1N1 vaccine (PANFLU.1), 15 micrograms per dose per 0.5 millilitre. Vaccines will be administered as a single 0.5 mL intramuscular injection in the deltoid muscle of the arm (randomized in one arm) at the first dose and the other arm for the second dose
  Arms: Group 2 : 15 μg pandemic influenza A/H1N1 vaccine
Biological: Seasonal trivalent vaccine — Trivalent Inactivated Influenza Vaccine (ANFLU), 7.5 micrograms of each strain per dose per 0.25 millilitre. Vaccines will be administered as a single 0.25 mL intramuscular injection in the deltoid muscle of the arm (randomized in one arm) at the first dose and the other arm for the second dose
  Arms: Group 3 : 7.5 μg seasonal trivalent vaccine

SUMMARY:
A single center, observer-masked, randomized clinical trial is to be conducted in 6-35 months infants to evaluate the safety and immunogenicity of Sinovac's influenza A/H1N1 Vaccine (PANFLU.1).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female aged between 6 and 35 months
2. Full-term birth, birth weight 2,500 grams or more
3. provided birth certification or vaccination card Parent(s) or legal guardian(s) are able to understand and sign the informed consent

Exclusion Criteria:

1. Cases, cured cases and close contact of influenza A (H1N1) virus
2. Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine, such as egg, egg protein, etc
3. Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain
4. Symptoms of acute infection within a week
5. Autoimmune disease or immunodeficiency
6. Congenital malformation, developmental disorders or serious chronic diseases (such as Down's syndrome, diabetes, sickle cell anemia or neurological disorders)
7. Asthma that is unstable or required emergent care, hospitalization or intubation during the past two years or that required the use of oral or intravenous corticosteroids
8. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
9. History or family history of convulsions, epilepsy, brain disease and psychiatric
10. Asplenia, functional asplenia or any condition resulting in the absence or removal o the spleen
11. Guillain-Barre Syndrome
12. Administration of 2009-2010 seasonal vaccine
13. History of any blood products within 3 months
14. Administration of any other investigational research agents within 30 days
15. Administration of any live attenuated vaccine within 30 days
16. Administration of subunit or inactivated vaccines within 14 days
17. Be receiving anti-TB prophylaxis or therapy currently
18. Axillary temperature > 37.0 centigrade at the time of dosing
19. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 310 (Actual)
Dates: Start 2009-12; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Evaluate immunogenicity of H1N1 vaccine with seasonal influenza vaccine in infants | 3 months

SECONDARY OUTCOMES:
Evaluate safety of H1N1 vaccine with seasonal influenza vaccine in infants | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- GuangXi Center for Diseases Control and Prevention, Guilin, Guangxi, China

REFERENCES:
- [Derived] Li YP, Li W, Liang XF, Liu Y, Huang XC, Li CG, Li RC, Wang JZ, Wang HQ, Yin WD. Immunogenicity and safety of a 2009 pandemic influenza A (H1N1) monovalent vaccine in Chinese infants aged 6-35 months: a randomized, double-blind, controlled phase I clinical trial. Influenza Other Respir Viruses. 2013 Nov;7(6):1297-307. doi: 10.1111/irv.12028. Epub 2012 Nov 8. PMID 23134570